CLINICAL TRIAL: NCT02334540
Title: Satiety Effects of Pulses Compared to Matched Protein Smoothie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 1412M57002
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Food Selection
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- purses or a calorie/protein matched smoothie (Other)
  Interventions: Dietary Supplement: purses; Dietary Supplement: a calorie/protein matched smoothie

INTERVENTIONS:
Dietary Supplement: purses — food intake
Dietary Supplement: a calorie/protein matched smoothie

SUMMARY:
The satiety effects of pulses compared to a matched smoothie will be measured.

DETAILED DESCRIPTION:
The investigators will compare satiety and food intake after consumption of purses or a calorie/protein matched smoothie

ELIGIBILITY:
Inclusion Criteria:

* healthy, normal body weight,

Exclusion Criteria:

* smoker, restrained eating habits, recent weight change, history of disease, vegetarian, do not normally eat breakfast or lunch, are pregnant or lactating, have irregular menstrual cycles

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
satiety | 120 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Food Science and Nutrition, Saint Paul, Minnesota, United States